CLINICAL TRIAL: NCT02579512
Title: Non Invasive Extra-corporeal ECG Signal Analysis Algorithm( NID Algorithm) for Myocardial Ischemia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Taichung Veterans General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: IGA1041203
Record Dates: First submitted 2015-07-13; First posted 2015-10-19 (Estimated); Last update posted 2015-10-19 (Estimated); Status verified 2015-09

CONDITIONS: Acute Coronary Syndrome; Myocardial Ischemia
MeSH Terms: conditions — Acute Coronary Syndrome; Myocardial Ischemia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- Extra-corporeal ECG Signal Analysis
  Interventions: Other: Extra-corporeal ECG signal analysis

INTERVENTIONS:
Other: Extra-corporeal ECG signal analysis — The NIA algorithm is similar to the traditional 12-lead ECG equipment. By analyzing patient data, NIA algorithm provides more detailed results compared to traditional 12-lead ECG. Patients with suspected coronary artery disease are conventionally diagnosed and treated by cardiac catheterization. However, cardiac catheterization is invasive procedure. Unless clinical diagnosis is evident before cardiac catheterization, a treadmill exercise test, a nuclear medicine myocardial perfusion test, or a multi-direction coronary CT angiogram is usually performed to increase the accuracy of diagnosis. But these examinations are not accessible to all patients, and are time-consuming and costly.

SUMMARY:
The NIA algorithm is similar to the traditional 12-lead ECG equipment. By analyzing patient data, NIA algorithm provides more detailed results compared to traditional 12-lead ECG. Patients with suspected coronary artery disease are conventionally diagnosed and treated by cardiac catheterization. However, cardiac catheterization is invasive procedure. Unless clinical diagnosis is evident before cardiac catheterization, a treadmill exercise test, a nuclear medicine myocardial perfusion test, or a multi-direction coronary CT angiogram is usually performed to increase the accuracy of diagnosis. But these examinations are not accessible to all patients, and are time-consuming and costly.

DETAILED DESCRIPTION:
In this project, the investigators hope to compare the data collected under this new technology of NIA algorithm with results from final diagnoses of cardiac catheterization. As the NIA algorithm is a fast and less costly, if it provides more sensitivity and specificity than does exercise ECG, nuclear myocardial perfusion test, and high-resolution coronary CT angiogram, it will expedite diagnosis for patients with coronary artery disease.

ELIGIBILITY:
Inclusion Criteria:

* patient with acute coronary syndrome who accepted percutaneous coronary intervention

Exclusion Criteria:

* no percutaneous coronary intervention

Ages: 20 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: myocardial Ischemia
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2015-06; Primary Completion 2016-05 (Estimated)

PRIMARY OUTCOMES:
Major Adverse Cardiac Events (MACE) | within the first 180 days after PCI (percutaneous coronary intervention)
  MACE including de novo lesion , intra-stent stenosis, cardiac death and re-myocardial infarction

CONTACTS AND LOCATIONS:
Locations (1):
- Taichung Veterans General Hospital, Taichung, Taiwan

REFERENCES:
- [Result] Lipton JA, Warren SG, Broce M, Abboud S, Beker A, Sornmo L, Lilly DR, Maynard C, Lucas BD Jr, Wagner GS. High-frequency QRS electrocardiogram analysis during exercise stress testing for detecting ischemia. Int J Cardiol. 2008 Feb 29;124(2):198-203. doi: 10.1016/j.ijcard.2007.02.002. Epub 2007 Apr 25. PMID 17462756
- [Result] Sharir T, Merzon K, Kruchin I, Bojko A, Toledo E, Asman A, Chouraqui P. Use of electrocardiographic depolarization abnormalities for detection of stress-induced ischemia as defined by myocardial perfusion imaging. Am J Cardiol. 2012 Mar 1;109(5):642-50. doi: 10.1016/j.amjcard.2011.10.022. Epub 2011 Dec 9. PMID 22169126
- [Result] Choi JO, Chang SA, Park SJ, Lee SC, Park SW. Improved detection of ischemic heart disease by combining high-frequency electrocardiogram analysis with exercise stress echocardiography. Korean Circ J. 2013 Oct;43(10):674-80. doi: 10.4070/kcj.2013.43.10.674. Epub 2013 Oct 30. PMID 24255651